CLINICAL TRIAL: NCT07297966
Title: Evaluation of the Clinical Efficacy of Antrrix Probiotics in Improving Recurrent Respiratory Infections in Infants and Young Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Min-Tze LIONG (Other)
Collaborators: Xinyi City People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Min-Tze LIONG, Prof., Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: (2024)-0001
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Respiratory Tract Infections
Keywords: RRTI; probiotic; RCT; children
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Daily 2 × 10 9 CFU per 6 drops containing Lactobacillus rhamnosus CRL1505+Bifidobacterium brevis M-16V strain in MCT oil
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Daily 6 drops of MCT oil without probiotic
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Daily 2 × 10 9 CFU per 6 drops containing Lactobacillus rhamnosus CRL1505+Bifidobacterium brevis M-16V strain in MCT oil
  Arms: Probiotic
Dietary Supplement: Placebo — Daily 6 drops MCT oil without probiotics
  Arms: Placebo

SUMMARY:
This study is an 8-weeks, randomized controlled trial involving children under 6 years of age who meet clinical diagnostic criteria for RRTI. Participants are randomized to receive either probiotic or placebo. The primary clinical outcomes assessed are duration and frequency of respiratory symptoms and quality of life. To investigate potential mechanisms, stool samples were collected pre- and post-intervention for 16S rRNA gene sequencing to analyze changes in gut microbiota composition and identify specific bacterial taxa associated with clinical improvements.

DETAILED DESCRIPTION:
Recurrent respiratory tract infection (RRTI) is a common pediatric condition with an increasing yearly incidence, seriously impacting children's growth, development, and quality of life. Younger children are particularly vulnerable, with notably high incidence rates in those under five years of age. RRTI can hinder physical development, contribute to the emergence of antibiotic resistance, increase school absenteeism, and place significant economic stress on families and the healthcare system. The underlying causes and disease mechanisms of RRTI are multifactorial, involving immune immaturity, environmental exposures, and microbial imbalance. Growing evidence suggests that disruptions in the gut microbiota may influence respiratory health through the gut-lung axis. Probiotics, by supporting microbiota homeostasis and modulating immune responses, have demonstrated potential in reducing the frequency and severity of respiratory infections in children. Given these connections, further investigation into the targeted use of probiotics to improve clinical outcomes in RRTI is essential for advancing preventive and therapeutic strategies in pediatric care.

Some pathways are proposed to explain how probiotics may improve recurrent respiratory tract infections (RRTI). The gastrointestinal tract and respiratory tract are interconnected components of the mucosal immune system. Immune responses generated in the gut can influence distant mucosal sites, including the lungs. Probiotics can stimulate gut-associated lymphoid tissue, leading to enhanced production of antigen-specific immunoglobulins (IgG, IgA), cytokines, and short-chain fatty acids. These immune mediators circulate systemically and contribute to strengthened respiratory defenses. In addition, the respiratory tract possesses its own microbial ecosystem, and maintaining the stability of this respiratory microbiota is essential for safeguarding respiratory health.

Children affected by RRTI often exhibit decreased levels of beneficial bacteria such as Bifidobacteria and Lactobacilli in the intestines. Dysbiosis weakens both local and systemic immunity, particularly through reduced production of immunoglobulins such as IgA. Probiotic supplementation can help restore microbial balance and enhance the host's immune profile. Reported outcomes include fewer and milder respiratory infections, shorter symptom duration, and improved immune parameters such as increased immunoglobulin levels and a more favorable T-cell profile. Importantly, probiotics have demonstrated a strong safety profile in pediatric populations.

Based on current scientific understanding, this project will focus on children under 6 years of age who meet clinical diagnostic criteria for RRTI. Probiotics, containing strains Dipro-CRL1505 and M-16V strains, will be administered for 8 weeks to evaluate clinical benefits and safety outcomes. Additionally, 16S rRNA sequencing will assess gut microbiota composition before treatment, at 4 weeks, and at 8 weeks. Through these combined clinical and microbiological measures, the study aims to clarify the therapeutic potential and underlying mechanisms of this probiotic intervention in children with RRTI.

ELIGIBILITY:
Inclusion Criteria:

* Age < 6 years, gender not limited;
* Meets the clinical diagnostic criteria for recurrent respiratory tract infections (Clinical Diagnosis and Treatment Pathway for Recurrent Respiratory Tract Infections in Children (2022 Edition) 10 );
* Parents or other legal guardians of the child fully understand the trial and voluntarily sign informed consent forms before the start of any research procedure;
* Willing to discontinue the use of other probiotics during the trial;
* Agree to the collection of fecal biological samples during this trial.

Exclusion Criteria:

* Those deemed by the investigator to have poor compliance or be unsuitable for participation;
* Allergic to the investigational product and its components;
* Allergic to respiratory tract infection drugs and their components;
* Respiratory infections caused by underlying diseases such as primary immunodeficiency diseases, acquired immunodeficiency syndrome (ADRS), congenital airway malformations, congenital heart disease, gastroesophageal reflux disease (GERD), and pulmonary dysplasia;
* Patients with severe malnutrition, rickets, and severe primary diseases of the heart, brain, liver, kidney, and hematopoietic systems;
* Use probiotic preparations, antibiotics, immunostimulants, or immunosuppressants 4 weeks before participating in the experiment.

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory symptoms in children upon administration of probiotic or placebo as assessed via clinical questionnaire | day 1, day 7, day 14, week 4, week 8
  Differences in severity of respiratory symptoms in children upon administration of probiotic or placebo, assessed using a hospital-based clinical questionnaire scored on a 5-point ordinal scale (0 = no symptoms to 4 = severe symptoms), with lower scores indicating better respiratory status.

SECONDARY OUTCOMES:
Quality of life in children upon administration of probiotic or placebo via clinical questionnaire | day 1, day 7, day 14, week 4, week 8
  Differences in quality of life in children upon administration of probiotic or placebo, assessed using a hospital-based caregiver-reported clinical questionnaire scored on a 5-point ordinal scale, with lower scores indicating better quality of life.
Microbiota profiles of fecal samples in young children upon administration of probiotic, lactulose or their combinations as assessed via 16s rRNA gene sequencing | day 1, day 7, day 14, week 4, week 8
  Differences in microbiota profiles in fecal sample of children upon administration of probiotic or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Sitao Li, MD., Principal Investigator — The Sixth Affiliated Hospital of Sun Yat-sen University, Xinyi People's Hospital
Locations (2):
- Xinyi City People's Hospital, Xingyi, Guangdong, China
- Universiti Sains Malaysia, George Town, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No